CLINICAL TRIAL: NCT01004432
Title: A Golimumab Phase 3b, Multicenter, Switch Assessment of Subcutaneous and Intravenous Efficacy in Rheumatoid Arthritis Patients Who Have Inadequate Disease Control Despite Treatment With Etanercept (ENBREL) or Adalimumab (HUMIRA)
Brief Title: Golimumab in Rheumatoid Arthritis Participants With an Inadequate Response to Etanercept (ENBREL) or Adalimumab (HUMIRA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Biotech, Inc. (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR016663; CNTO148ART3002 (Other: Janssen Biotech Inc.); 2009-010582-23 (EudraCT Number); GO SAVE (Other: Janssen Biotech Inc.)
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Results first posted 2014-05-13 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Arthritis; Arthritis, Rheumatoid; Autoimmune Diseases
Keywords: humira, remicade; rheumatoid arthritis; enbrel failure; humira failure; arthritis; enbrel
MeSH Terms: conditions — Arthritis; Arthritis, Rheumatoid; Autoimmune Diseases | interventions — golimumab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Open-label (OL) Overall Group: Golimumab 50 mg SC + MTX (Experimental): All enrolled and dosed participants receive golimumab 50 milligram (mg) subcutaneous (SC) injection every 4 weeks + Methotrexate (MTX) from Week 0 to Week 12.
  Interventions: Drug: Golimumab 50 mg SC; Drug: Methotrexate (MTX)
- Double blind (DB) Group 2a: Golimumab 50mg SC & Placebo IV+MTX (Experimental): Participants, who do not achieve Disease Activity Score in 28 joints (DAS28) good response at Week 16, will be randomly assigned to receive golimumab 50 mg SC injection every 4 weeks + MTX from Week 16 to Week 48, along with placebo matched to golimumab intravenous infusion (IV) at Week 16, 20, 28, 36, and 44.
  Interventions: Drug: Golimumab 50 mg SC; Drug: Methotrexate (MTX); Drug: Placebo IV
- DB Group 2b: Golimumab 2mg/kg IV & Placebo SC + MTX (Experimental): Participants, who do not achieve DAS28 good response at Week 16, will be randomly assigned to receive golimumab 2 milligram per kilogram (mg/kg) intravenous infusion (IV) + MTX, at Week 16, 20, 28, 36 and 44, along with placebo matched to golimumab SC injection every 4 weeks from Week 16 to Week 48.
  Interventions: Drug: Golimumab 2 mg/kg IV; Drug: Methotrexate (MTX); Drug: Placebo SC
- OL Group 1: Golimumab 50 mg SC + MTX (Experimental): Participants, who achieve DAS28 good response at Week 16, will receive golimumab 50 mg SC injection every 4 weeks + MTX from Week 16 to Week 48.
  Interventions: Drug: Golimumab 50 mg SC; Drug: Methotrexate (MTX)
- OL Study Extension Group: Golimumab 50 mg SC + MTX (Experimental): Participants who complete the main study (Week 0 to Week 52), do not meet lack of efficacy criteria, and participate in the OL study extension, will receive golimumab 50 mg SC injection every 4 weeks + MTX from Week 52 to Week 72.
  Interventions: Drug: Golimumab 50 mg SC; Drug: Methotrexate (MTX)

INTERVENTIONS:
Drug: Golimumab 50 mg SC — Golimumab 50 milligram (mg) subcutaneous (SC) injection every 4 weeks.
  Arms: Double blind (DB) Group 2a: Golimumab 50mg SC & Placebo IV+MTX; OL Group 1: Golimumab 50 mg SC + MTX; OL Study Extension Group: Golimumab 50 mg SC + MTX; Open-label (OL) Overall Group: Golimumab 50 mg SC + MTX
Drug: Golimumab 2 mg/kg IV — Golimumab 2 milligram per kilogram (mg/kg) intravenous infusion every 8 weeks.
  Arms: DB Group 2b: Golimumab 2mg/kg IV & Placebo SC + MTX
Drug: Methotrexate (MTX) — Participants will continue taking their current Methotrexate (MTX) treatment regimen.
Drug: Placebo SC — Placebo matched to golimumab SC injection every 4 weeks.
  Arms: DB Group 2b: Golimumab 2mg/kg IV & Placebo SC + MTX
Drug: Placebo IV — Placebo matched to golimumab intravenous infusion every 8 weeks.
  Arms: Double blind (DB) Group 2a: Golimumab 50mg SC & Placebo IV+MTX

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of switching rheumatoid arthritis (RA) participants who have an inadequate response to their current treatment with either etanercept + methotrexate or adalimumab + methotrexate to treatment with golimumab 50 milligram (mg) subcutaneous (SC) injection (a needle inserted under the skin in the back of upper arm, upper thigh or stomach area) every 4 weeks + methotrexate. This study is also designed to evaluate the benefit and safety of switching participants from treatment with golimumab 50 mg subcutaneous injection every 4 weeks + methotrexate to golimumab 2 milligram per kilogram (mg/kg) intravenous every 8 weeks + methotrexate, for those who do not achieve a marked improvement of their RA at Week 16.

DETAILED DESCRIPTION:
The study consists of a main study and a voluntary, open-label (participants and researchers are aware about the treatment participants are receiving), 24-week study extension. The main study includes a Screening Run-in Period (Week -6 to Week 0), an Open-label Treatment Period (Week 0 to Week 16), an Open-label or Double-blind Treatment Period (Week 16 to Week 52). The main study also includes a Follow-up Period from Week 52 through Week 64 for those participants who will not participate in the 24-week study extension. Participants, participating in 24-week extension (at Week 52), will receive open-label golimumab SC injections every 4 weeks from Week 52 up to Week 72 and will be followed-up up to Week 88. All eligible participants will initiate the treatment with open-label golimumab SC injection every 4 weeks up to Week 12. At Week 16, depending upon the treatment response either participants will continue to receive open-label golimumab SC injection every 4 weeks up to Week 48 or participants will be randomly assigned to receive following 2 treatments: 1- golimumab 50mg SC injection every 4 weeks along with placebo intravenous infusion every 8 weeks through Week 48; 2- Placebo SC injection every 4 weeks along with golimumab 2mg/kg intravenous infusion every 8 weeks through Week 48. At Week 52, participants who choose to participate in the 24-week study extension will receive open-label golimumab 50 mg SC injections every 4 weeks through Week 72. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Have inadequate RA disease control prior to the first administration of study agent despite treatment with etanercept (Enbrel) + methotrexate or adalimumab (Humira) + methotrexate (MTX)
* Must have received a stable dose of MTX greater than or equal to (>=) 7.5 milligram (mg) per week to less than or equal to (<=) 25 mg per week for at least 4 consecutive weeks prior to the first screening visit and must plan to maintain that dose throughout the study
* Participants must have received etanercept or adalimumab in combination with MTX for a minimum of 3 months prior to the first visit
* Negative tuberculosis (TB) test
* Are capable of providing informed consent, which must be obtained prior to any study-related procedures

Exclusion Criteria:

* Have a history of latent or active granulomatous infection, including TB, histoplasmosis, or coccidioidomycosis, or are frequently in contact with individuals who carry active TB infection
* Have inflammatory diseases other than RA, including but not limited to psoriatic arthritis, ankylosing spondylitis, systemic lupus erythematosus, primary Sjogren's or Lyme disease
* Have demonstrated a discernible improvement in disease activity between screening and prior to the first golimumab injection at Week 0
* Have any known malignancy or have a history of malignancy within the previous 5 years (with the exception of a nonmelanoma skin cancer that has been treated with no evidence of recurrence)
* Have a history of lymphoproliferative disease, including lymphoma, or signs and symptoms suggestive of possible lymphoproliferative disease such as lymphadenopathy of unusual size or location

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 433 (Actual)
Dates: Start 2009-12; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Biotech, Inc. Clinical Trial, Study Director — Janssen Biotech, Inc.
Locations (117):
- United States (89):
  - Birmingham, Alabama
  - Huntsville, Alabama
  - Tuscaloosa, Alabama
  - Mesa, Arizona
  - Phoenix, Arizona
  - Hot Springs, Arkansas
  - Little Rock, Arkansas
  - Covina, California
  - Hemet, California
  - Loma Linda, California
  - Long Beach, California
  - Murrieta, California
  - Santa Maria, California
  - Santa Monica, California
  - Torrance, California
  - Van Nuys, California
  - Victorville, California
  - Whittier, California
  - Bridgeport, Connecticut
  - Hamden, Connecticut
  - Trumbull, Connecticut
  - Aventura, Florida
  - Fort Lauderdale, Florida
  - Jacksonville, Florida
  - Naples, Florida
  - Orange Park, Florida
  - Orlando, Florida
  - Palm Harbor, Florida
  - Plantation, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Duluth, Georgia
  - Coeur d'Alene, Idaho
  - Idaho Falls, Idaho
  - Rockford, Illinois
  - South Bend, Indiana
  - Bettendorf, Iowa
  - Kansas City, Kansas
  - Bowling Green, Kentucky
  - Monroe, Louisiana
  - New Orleans, Louisiana
  - Wheaton, Maryland
  - Rochester, Minnesota
  - Flowood, Mississippi
  - Tupelo, Mississippi
  - Clayton, Missouri
  - Florissant, Missouri
  - Lincoln, Nebraska
  - Freehold, New Jersey
  - Brooklyn, New York
  - Mineola, New York
  - Plainview, New York
  - Rochester, New York
  - Smithtown, New York
  - Charlotte, North Carolina
  - Greenville, North Carolina
  - Hickory, North Carolina
  - Wilmington, North Carolina
  - Akron, Ohio
  - Columbus, Ohio
  - Mayfield, Ohio
  - Middleburg Heights, Ohio
  - Edmond, Oklahoma
  - Oklahoma City, Oklahoma
  - Lake Oswego, Oregon
  - Bethlehem, Pennsylvania
  - Duncansville, Pennsylvania
  - West Reading, Pennsylvania
  - Wexford, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Myrtle Beach, South Carolina
  - Hixson, Tennessee
  - Jackson, Tennessee
  - Kingsport, Tennessee
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - Carrollton, Texas
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Arlington, Virginia
  - Chesapeake, Virginia
  - Seattle, Washington
  - Spokane, Washington
  - Beckley, West Virginia
  - Clarksburg, West Virginia
  - Glendale, Wisconsin
- Vienna, Austria
- Belgium (5):
  - Brussels
  - Genk
  - Ghent
  - Liège
  - Merksem
- Canada (8):
  - Edmonton, Alberta
  - Kelowna, British Columbia
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Hamilton, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - St. Johns
- Germany (4):
  - Hamburg
  - Herne
  - München
  - Ratingen
- Greece (2):
  - Heraklion- Crete
  - Thessalonikis
- Stockholm, Sweden
- United Kingdom (7):
  - Cannock
  - Leeds
  - London
  - Manchester
  - Merseyside
  - Newcastle upon Tyne
  - Wigan

REFERENCES:
- [Derived] Dehoratius RJ, Brent LH, Curtis JR, Ellis LA, Tang KL. Satisfaction with Subcutaneous Golimumab and its Auto-Injector among Rheumatoid Arthritis Patients with Inadequate Response to Adalimumab or Etanercept. Patient. 2018 Jun;11(3):361-369. doi: 10.1007/s40271-018-0297-5. PMID 29427176
- [Derived] Huffstutter JE, Kafka S, Brent LH, Matucci-Cerinic M, Tang KL, Chevrier M, Sprabery T, DeHoratius RJ. Clinical response to golimumab in rheumatoid arthritis patients who were receiving etanercept or adalimumab: results of a multicenter active treatment study. Curr Med Res Opin. 2017 Apr;33(4):657-666. doi: 10.1080/03007995.2016.1277195. Epub 2017 Jan 25. PMID 28035867

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-label (OL) Overall Group: Golimumab 50 mg SC + MTX: All enrolled and dosed participants received golimumab 50 mg SC injection every 4 weeks + MTX from Week 0 to Week 12.
- OL Group 1: Golimumab 50 mg SC + MTX: Participants, who achieved Disease Activity Score in 28 joints (DAS28) good response at Week 16, received Golimumab 50 milligram (mg) subcutaneous (SC) injection every 4 weeks + Methotrexate (MTX) from Week 16 to Week 48.
- Double Blind (DB) Group 2a: Golimumab 50mg SC & Placebo IV+MTX: Participants, who did not achieve DAS28 good response at Week 16, were randomly assigned to receive golimumab 50 mg SC injection every 4 weeks + MTX from Week 16 to Week 48, along with placebo matched to golimumab intravenous infusion (IV) at Week 16, 20, 28, 36, and 44.
- DB Group 2b: Golimumab 2mg/kg IV & Placebo SC + MTX: Participants, who did not achieve DAS28 good response at Week 16, were randomly assigned to receive golimumab 2 milligram per kilogram (mg/kg) intravenous infusion (IV) + MTX, at Week 16, 20, 28, 36 and 44, along with placebo matched to golimumab SC injection every 4 weeks from Week 16 to Week 48.
- OL Study Extension Group: Golimumab 50 mg SC + MTX: Participants who completed the main study (Week 0 to Week 52), not met lack of efficacy criteria, and participated in the OL study extension, received golimumab 50 mg SC injection every 4 weeks + MTX from Week 52 to Week 72.
Period: Open-label (OL) Period (Week 0 - 16)
Arm/Group | Open-label (OL) Overall Group: Golimumab 50 mg SC + MTX | OL Group 1: Golimumab 50 mg SC + MTX | Double Blind (DB) Group 2a: Golimumab 50mg SC & Placebo IV+MTX | DB Group 2b: Golimumab 2mg/kg IV & Placebo SC + MTX | OL Study Extension Group: Golimumab 50 mg SC + MTX
Started | 433 | 0 | 0 | 0 | 0
Completed | 350 (1 Participant died after completing open-label period. Discontinuation was noted as adverse event.) | 0 | 0 | 0 | 0
Not Completed | 83 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 20 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 29 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 17 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 15 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0 | 0
Period: OL/Double-Blind (DB) Period (Week 16-52)
Arm/Group | Open-label (OL) Overall Group: Golimumab 50 mg SC + MTX | OL Group 1: Golimumab 50 mg SC + MTX | Double Blind (DB) Group 2a: Golimumab 50mg SC & Placebo IV+MTX | DB Group 2b: Golimumab 2mg/kg IV & Placebo SC + MTX | OL Study Extension Group: Golimumab 50 mg SC + MTX
Started | 0 | 75 | 91 | 184 | 0
Completed | 0 | 65 | 54 | 126 | 0
Not Completed | 0 | 10 | 37 | 58 | 0
Not completed — Adverse Event | 0 | 1 | 5 | 6 | 0
Not completed — Protocol Violation | 0 | 3 | 3 | 4 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 4 | 7 | 0
Not completed — Death | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 2 | 24 | 37 | 0
Not completed — Lost to Follow-up | 0 | 3 | 1 | 3 | 0
Period: OL Study Extension (Week 52 - 76)
Arm/Group | Open-label (OL) Overall Group: Golimumab 50 mg SC + MTX | OL Group 1: Golimumab 50 mg SC + MTX | Double Blind (DB) Group 2a: Golimumab 50mg SC & Placebo IV+MTX | DB Group 2b: Golimumab 2mg/kg IV & Placebo SC + MTX | OL Study Extension Group: Golimumab 50 mg SC + MTX
Started | 0 | 0 | 0 | 0 | 212
Completed | 0 | 0 | 0 | 0 | 194
Not Completed | 0 | 0 | 0 | 0 | 18
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 10

BASELINE CHARACTERISTICS:
Groups:
- OL Overall Group: Golimumab 50 mg SC + MTX: All enrolled and dosed participants received golimumab 50 mg SC injection every 4 weeks + MTX from Week 0 to Week 12.
Arm/Group | OL Overall Group: Golimumab 50 mg SC + MTX
Number analyzed (Participants) | 433
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (11.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 358
  Male | 75
Region of Enrollment [Number; unit: participants]
  Austria | 1
  Belgium | 9
  Canada | 37
  Germany | 7
  Greece | 8
  Italy | 12
  Sweden | 1
  United Kingdom | 9
  United States | 349

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Erythrocyte Sedimentation Rate (ESR)-Based American College of Rheumatology [ACR] 20 Response at Week 14
Description: Erythrocyte Sedimentation Rate (ESR)-based ACR 20 response: greater than or equal to (>=) 20 percent (%) improvement from Baseline in tender (68 joints assessed) and swollen (66 joints assessed) joint counts and >=20% improvement from Baseline in 3 of the following 5 assessments: 1- Participant's assessment of pain using Visual Analog Scale (VAS) (0 to 10 centimeters [cm]), 2- Participant's global assessment of disease activity using VAS (0 to 10 cm), 3- Physician's global assessment of disease activity using VAS (0 to 10 cm), 4- Participant's assessment of physical function as measured by the Disability Index of the Health Assessment Questionnaire (HAQ-DI) (score of 0-3 in 8 functional areas), 5- ESR.
Time Frame: Week 14
Population: Modified Intent To Treat (mITT) population included all enrolled participants who had Week 0 measurements and received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OL Overall Group: Golimumab 50 mg SC + MTX
Number analyzed (Participants) | 433
percentage of participants | 34.9 [30.4 to 39.4]
Statistical Analysis 1: Comparison: OL Overall Group: Golimumab 50 mg SC + MTX; null hypothesis: proportion <=0.2; Test type: Superiority or Other; p < 0.0001, Chi-squared — One sided test adjusting for conducting one interim analysis; Percentage achive ACR 20 response = 34.9, 95% CI 2-sided [30.4 to 39.4]

2. Secondary Outcome: Percentage of Participants Who Achieved Erythrocyte Sedimentation Rate (ESR)-Based ACR20 Response at Week 2
Description: as for outcome 1
Time Frame: Within 2 weeks of initiating therapy
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OL Overall Group: Golimumab 50 mg SC + MTX
Number analyzed (Participants) | 433
percentage of participants | 24.5 [20.4 to 28.5]

3. Secondary Outcome: Percentage of Participants Who Achieved Erythrocyte Sedimentation Rate (ESR)-Based Disease Activity Score (DAS28) Response at Week 16 and Maintained Response Through Week 52
Description: Erythrocyte Sedimentation Rate (ESR)-based disease activity score for 28-joints count (DAS28) as defined by European League Against Rheumatism (EULAR), response criteria was used to assess individual response as none, moderate, or good, depending on the extent of change from Baseline and the level of disease activity reached. A participant was classified as having achieved a DAS28 good response if, DAS28 was less than or equal to (<=) 3.2 at a given visit and improvement from Baseline was >1.2. Percentage of participants, who achieved ESR-based DAS 28 good response at Week 16 and maintained that response through Week 52, is reported.
Time Frame: Week 52
Population: Open-label modified Intent To Treat (mITT) population included all participants, who received at least 1 open-label golimumab 50 mg SC injection during the continued open-label/ double-blind treatment period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OL Group 1: Golimumab 50 mg SC + MTX
Number analyzed (Participants) | 75
percentage of participants | 22.7 [13.2 to 32.1]

4. Secondary Outcome: Percentage of Participants Who Achieved Erythrocyte Sedimentation Rate (ESR)-Based ACR20 Response at Week 52 Relative to Week 16
Description: Erythrocyte Sedimentation Rate (ESR)-based ACR 20 response: >=20 % improvement from Week 16 in tender (68 joints assessed) and swollen (66 joints assessed) joint counts and >=20% improvement from Week 16 in 3 of the following 5 assessments: 1- Participant's assessment of pain using VAS (0 to 10 cm), 2- Participant's global assessment of disease activity using VAS (0 to 10 cm), 3- Physician's global assessment of disease activity using VAS (0 to 10 cm), 4- Participant's assessment of physical function as measured by the Disability Index of the Health Assessment Questionnaire (HAQ-DI) (score of 0-3 in 8 functional areas), 5- ESR. Percentage of participants, who achieved ESR-based ACR 20 responses at Week 52 relative to Week 16, is reported.
Time Frame: Week 52
Population: Double-blind modified Intent To Treat (mITT) population included participants who were randomized at Week 16 to SC or IV golimumab (Groups 2a and 2b) and received at least 1 dose of study drug after randomization.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- DB Group 2a: Golimumab 50 mg SC & Placebo IV + MTX: Participants, who did not achieved DAS28 good response at Week 16, were randomly assigned to receive golimumab 50 mg SC injection every 4 weeks + MTX from Week 16 to Week 48, along with placebo matched to golimumab intravenous infusion (IV) at Week 16, 20, 28, 36, and 44.
- DB Group 2b: Golimumab 2 mg/kg IV & Placebo SC + MTX: Participants, who did not achieve DAS28 good response at Week 16, were randomly assigned to receive golimumab 2 milligram per kilogram (mg/kg) intravenous infusion (IV) + MTX, at Week 16, 20, 28, 36 and 44, along with placebo matched to golimumab SC injection every 4 weeks from Week 16 to Week 48.
Arm/Group | DB Group 2a: Golimumab 50 mg SC & Placebo IV + MTX | DB Group 2b: Golimumab 2 mg/kg IV & Placebo SC + MTX
Number analyzed (Participants) | 91 | 184
percentage of participants | 13.2 [6.2 to 20.1] | 9.2 [5.1 to 13.4]

5. Secondary Outcome: Percentage of Participants Who Achieved ESR-based and C-Reactive Protein (CRP)-Based ACR20 Response at Week 76 Relative to Week 16
Description: Erythrocyte Sedimentation Rate (ESR)-based/ C Reactive Protein (CRP)-based ACR 20 response: >=20 % improvement from Week 16 in tender (68 joints assessed) and swollen (66 joints assessed) joint counts and >=20% improvement from Week 16 in 3 of the following 5 assessments: 1- Participant's assessment of pain using VAS (0 to 10 cm), 2- Participant's global assessment of disease activity using VAS (0 to 10 cm), 3- Physician's global assessment of disease activity using VAS (0 to 10 cm), 4- Participant's assessment of physical function as measured by the Disability Index of the Health Assessment Questionnaire (HAQ-DI) (score of 0-3 in 8 functional areas), 5- ESR or CRP. Percentage of participants, who achieved ESR/ CRP-based ACR 20 responses at Week 76 relative to Week 16, is reported.
Time Frame: Week 76
Population: Study extension mITT population included all participants, who were enrolled into the 24-week study extension period at Week 52, and received at least 1 golimumab SC injection during the study extension period. Participants reported in other groups are subgroups of 'Study Extension OL Group' by treatment received in the OL/DB phase (Weeks 16-52).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | OL Group 1: Golimumab 50 mg SC + MTX | DB Group 2a: Golimumab 50 mg SC & Placebo IV + MTX | DB Group 2b: Golimumab 2 mg/kg IV & Placebo SC + MTX | OL Study Extension Group: Golimumab 50 mg SC + MTX
Number analyzed (Participants) | 63 | 47 | 102 | 212
percentage of participants
  ESR-based ACR 20 Response | 7.9 [1.3 to 14.6] | 8.5 [0.5 to 16.5] | 15.7 [8.6 to 22.7] | 11.8 [7.5 to 16.1]
  CRP-based ACR 20 Response | 7.9 [1.3 to 14.6] | 8.5 [0.5 to 16.5] | 17.6 [10.2 to 25.0] | 12.7 [8.2 to 17.2]

6. Secondary Outcome: Change in ESR-based DAS28 Score at Week 76 Relative to Week 52
Description: Erythrocyte Sedimentation Rate (ESR)-based disease activity score for 28-joints count (DAS28) was calculated from number of swollen joint counts (SJC) and tender joint counts (TJC) using 28 joints count, ESR, and patient global assessment of disease activity (participant rated arthritis activity assessment with scores ranging 0 to 10; higher scores indicated greater disease activity). Total ESR-based DAS28 score range: 0 to 9.4, higher score=more disease activity.
Time Frame: Week 52, 76
Population: Study extension mITT population. Here 'N' (number of participants analyzed) = participants evaluable for this measure and 'n' = participants evaluable at specified time point for each arm, respectively. Participants reported in other groups are subgroups of 'Study Extension OL Group' by treatment received in the OL/DB phase (Weeks 16-52).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OL Group 1: Golimumab 50 mg SC + MTX | DB Group 2a: Golimumab 50 mg SC & Placebo IV + MTX | DB Group 2b: Golimumab 2 mg/kg IV & Placebo SC + MTX | OL Study Extension Group: Golimumab 50 mg SC + MTX
Number analyzed (Participants) | 61 | 40 | 95 | 196
units on a scale
  Week 52 (n = 61, 40, 95, 196) | 3.182 (1.1109) [1.3 to 14.6] | 4.070 (0.8037) [0.5 to 16.5] | 4.394 (1.2389) [8.6 to 22.7] | 3.950 (1.2379) [7.5 to 16.1]
  Change at Week 76 (n = 57, 33, 84, 174) | -0.136 (1.2095) [1.3 to 14.6] | 0.209 (1.2253) [0.5 to 16.5] | -0.017 (1.0518) [10.2 to 25.0] | -0.013 (1.1386) [8.2 to 17.2]

ADVERSE EVENTS:
Arm/Group | OL Overall Group: Golimumab 50 mg SC + MTX | OL Group 1: Golimumab 50 mg SC + MTX | Double Blind (DB) Group 2a: Golimumab 50mg SC & Placebo IV+MTX | DB Group 2b: Golimumab 2mg/kg IV & Placebo SC + MTX | OL Study Extension Group: Golimumab 50 mg SC + MTX
Serious Adverse Events (participants affected / at risk) | 20/433 | 2/75 | 4/91 | 10/184 | 10/212
Other Adverse Events (participants affected / at risk) | 123/433 | 21/75 | 30/91 | 54/184 | 61/212
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OL Overall Group: Golimumab 50 mg SC + MTX (N=433) | OL Group 1: Golimumab 50 mg SC + MTX (N=75) | Double Blind (DB) Group 2a: Golimumab 50mg SC & Placebo IV+MTX (N=91) | DB Group 2b: Golimumab 2mg/kg IV & Placebo SC + MTX (N=184) | OL Study Extension Group: Golimumab 50 mg SC + MTX (N=212)
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1 | 1
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 2 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Wound infection staphylococcal (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Carotid artery occlusion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Intracranial aneurysm (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Polyneuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 1 | 0 | 0 | 3 | 1
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 1
Hepatitis C (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Breast cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OL Overall Group: Golimumab 50 mg SC + MTX (N=433) | OL Group 1: Golimumab 50 mg SC + MTX (N=75) | Double Blind (DB) Group 2a: Golimumab 50mg SC & Placebo IV+MTX (N=91) | DB Group 2b: Golimumab 2mg/kg IV & Placebo SC + MTX (N=184) | OL Study Extension Group: Golimumab 50 mg SC + MTX (N=212)
Bronchitis (Infections and infestations) | 12 | 2 | 6 | 11 | 4
Sinusitis (Infections and infestations) | 17 | 4 | 4 | 13 | 12
Upper respiratory tract infection (Infections and infestations) | 29 | 7 | 5 | 15 | 13
Urinary tract infection (Infections and infestations) | 24 | 3 | 2 | 11 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 20 | 2 | 8 | 8 | 11
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 13 | 2 | 9 | 9 | 11
Headache (Nervous system disorders) | 24 | 0 | 1 | 5 | 3
Depression (Psychiatric disorders) | 7 | 4 | 3 | 2 | 5

LIMITATIONS AND CAVEATS:
Since participants assigned to the double blind groups were non-responders to at least 2 anti-Tumor Necrosis Factors (TNF), thus comprising a very difficult group to treat.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days